CLINICAL TRIAL: NCT01357343
Title: Effect of an Integrative Approach of Chiropractic and Traditional Chinese Medicine Care on Low Back Pain: A Randomized Controlled Trial
Brief Title: Integrated Chiropractic and Acupuncture Treatment for Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Principal Investigator, Anupama KizhakkeVeettil, Assistant Professor, Southern California University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIZH003
Record Dates: First submitted 2011-03-22; First posted 2011-05-20 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Chiropractic; Acupuncture; Integrated care
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Chiropractic; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture (Active Comparator): Acupuncture needling, moxa, Tui Na and cupping
  Interventions: Other: Acupuncture
- Chiropractic care (Active Comparator): Chiropractic adjustments and active and passive physical modalities.
  Interventions: Other: Chiropractic
- Integrated Chiropractic and Acupuncture (Active Comparator)
  Interventions: Other: Chiropractic; Other: Acupuncture

INTERVENTIONS:
Other: Chiropractic — Spinal manipulation and active and passive therapy.
  Arms: Chiropractic care; Integrated Chiropractic and Acupuncture
Other: Acupuncture — Acupuncture needling, moxa, Tui Na and cupping.
  Arms: Acupuncture; Integrated Chiropractic and Acupuncture

SUMMARY:
This study is being conducted to compare the effectiveness of integrated chiropractic and acupuncture care for the management of low back pain.

DETAILED DESCRIPTION:
This study is being conducted at the Southern California University of Health Sciences. Eligible subjects will be randomized to one of three treatment groups: chiropractic care alone, acupuncture care alone, and chiropractic and acupuncture care combined.

Subjects will be treated on pragmatic basis for 60 days and then followed up for an additional 60 days. All examinations and treatments will be provided free of charge. The expected benefits for the participants are decreased pain and improved function.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older
* Have a current episode of low back pain

Exclusion Criteria:

* Received chiropractic treatment or other manipulative therapies within the last month
* Received acupuncture treatment within the last month
* Visceral, systemic or joint inflammatory disease with referred pain to the back or pelvis
* Non-mechanical low back pain
* A history of low back surgery
* Osteoporosis
* Spondylolisthesis
* Coagulation disorder or are taking anticoagulant medication
* Prolonged systemic corticosteroid medication
* Progressive unilateral lower limb muscle weakness
* Symptoms or signs of cauda equina syndrome (e.g., bowel or bladder dysfunction)
* Severe concurrent illness (e.g., cancer, heart diseases, psychiatric disorders)
* Known pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain numeric rating scale. | Change from baseline to 60 days
  This outcome will measure changes in the participant's level of low back pain.
Disability due to low back pain | Change from baseline to 60 days
  We will be using Roland-Morris scale to measure disability due to low back pain.

SECONDARY OUTCOMES:
Quality of life | Change from baseline to 60 days days
  Quality of life is often reduced due to low back pain. The SF-36 outcome measure will be used to determine if the treatment has any effect on quality of life of the participants.
Patient satisfaction with treatment | Change from baseline to 60 days
  We will be using Cherkin-satisfaction scale to measure patient's satisfaction with the treatment offered.
Self generated survey of outcomes | Change from baseline to 60 days days
  Frequency of symptoms, Medication use, Lost work time, Health services utilization

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Kizhakkeveettil, MAOM, Principal Investigator — Southern California University of Health Sciences
Locations (1):
- Southern California University of Health Sciences, Whittier, California, United States

REFERENCES:
- [Derived] Kizhakkeveettil A, Rose KA, Kadar GE, Hurwitz EL. Integrative Acupuncture and Spinal Manipulative Therapy Versus Either Alone for Low Back Pain: A Randomized Controlled Trial Feasibility Study. J Manipulative Physiol Ther. 2017 Mar-Apr;40(3):201-213. doi: 10.1016/j.jmpt.2017.01.002. Epub 2017 Mar 1. PMID 28259496